CLINICAL TRIAL: NCT07289191
Title: Design of tSCS Strategies to Promote Neural Plasticity and Improve Functional Outcomes During Rehabilitation of Locomotion
Brief Title: Development of a Novel Strategy to Analyze the Effect on Gait Using Transcutaneous Spinal Current Stimulation in Incomplete Spinal Cord Injured Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Guttmann (Other)
Responsible Party: Principal Investigator, Hatice Kumru, Principal Investigator, Institut Guttmann
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2.022.386
Record Dates: First submitted 2024-09-21; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries; Non Invasive Spinal Stimulation; Gait Disorders, Neurologic; Motor Function; Retardation; Stimulation Charecteristic
MeSH Terms: conditions — Spinal Cord Injuries; Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multisegmental tSCS combined with gait rehabilitation (Experimental)
  Interventions: Device: transcutaneous spinal cord stimulation
- Gait rehabilitation (Other): baseline, during transcutaneous spinal cord stimulation (tSCS) at C5, L1, Coc1, or combinations of two segments or multisegment stimulation, and the final assessment.
  Interventions: Device: transcutaneous spinal cord stimulation

INTERVENTIONS:
Device: transcutaneous spinal cord stimulation — This study consisted of: (i) baseline condition; and (ii) tSCS conditions: which consisted of 7 different combinations applied to different segments of the spinal cord in the randomized order: C5, L1, Coc1, C5+L1, C5+Coc1, L1+Coc1, C5+L1+Coc1 and than (iii) final condition: Individuals with SCI realized all clinical assessment after the last condition of tDCSs. We included the final control condition to ensure the reliability of our findings.
  Baseline, tSCSs, and final control conditions were conducted as part of three assessments: the 6MWT and MVC-QM and MVC-TA, Hmax/Mmax ratio.

SUMMARY:
To determine whether the combination of non-invasive spinal cord stimulation together with gait rehabilitation reduces spasticity and facilitates recovery of lower limb motor strength and gait function in patients with incomplete SCI, as well as studying the underlying physiopathological changes following incomplete SCI and its modulation by non-invasive stimulation techniques.

DETAILED DESCRIPTION:
Methodology: This task will involve the clinical and functional assessment of patients completing gait training with and without tSCS as defined in T4.2 to demonstrate the effects of tSCS and define the most favorable parameters. During this task, the assessments that will be completed will be defined by IG and then carried out according to the methodology that is set and agreed upon. Assessments will need to evaluate several factors:

* The American Spinal Cord Injury Association Impairment Scale (ASIA) and the International Standards for Neurological Classification of Spinal Cord Injury (ISNSCI)38 will be used to determine level and severity of SCI and to evaluate sensory and motor deficit.
* For gait outcome measures, 10 meters walking test (10MWT) and Walking Index for SCI (WISCI) II will be assessed.
* For spasticity evaluation, Modified Ashworth modified score (MAS) will be used.
* Neurophysiological studies may be included to study: 1) spinal cord excitability using F and H wave, 2) corticospinal conduction using transcraneal magnetic stimulation for MEP recording, and 3) muscle activity using surface EMG recording of lower limb muscles.

ELIGIBILITY:
Inclusion Criteria:

* Male or female more than 18 years old;
* With a stable traumatic o nor traumatic incomplete motor cervical or thoracic SCI;
* Time since SCI more than 6 months;
* American Spinal Injury Association Impairment Scale (AIS)-D who could realize gait at least 6 meters with or without technical help;
* Capacity for compression the nature of the study and signed informed consent.

Exclusion Criteria:

* Unstable medical condition (cancer, acute infections, etc.);
* Severe spasticity (≥ 3 score on the Modified Ashworth scale (MAS)),
* Peripheral nerve affectation;
* Ulcers on the electrode applied area;
* Intolerance of tSCS.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
6MWT | Baseline, after 3 weeks, and 1 week follow-up
  6 METER WALKING TEST

SECONDARY OUTCOMES:
MVC | Baseline, after 3 weeks, and 1 week follow-up
  Maximum voluntary contraction
Hmax\Max ratio | Baseline, after 3 weeks, and 1 week follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Guttmann, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No